CLINICAL TRIAL: NCT02900846
Title: Usefulness of Colour Doppler Flow Imaging in the Management of Lacrimal Gland Lesions
Brief Title: Colour Doppler Flow Imaging in Lacrimal Gland Lesions
Acronym: GLIR
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_ALR_2015_1
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Lacrimal Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Retrospective medical charts and medical imaging files review of patients suffering from lacrimal fossa lesions who underwent ocular ultrasonography with color flow doppler imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from lacrimal fossa tumor
* Orbital ultrasonography performed, including doppler flow imaging
* Histopathological characterization of the tumor obtained after surgical removal

Exclusion Criteria:

* Absence of histopathological characterization
* Absence of documented ultrasound doppler flow imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from lacrimal fossa tumors explored with ultrasonography including doppler flow imaging
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2003-01; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pulsed wave doppler resistance index in tumor vascularization | 1 week